CLINICAL TRIAL: NCT00404365
Title: Maximizing Utilization of Depression Screening in Lung Cancer Patients: A Randomized Trial
Brief Title: Depression Screening in Patients With Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Lucille P. Markey Cancer Center at University of Kentucky (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Mskcc 06-038; R01CA115349 (NIH); P30CA008748 (NIH); MSKCC-06038; NCT00369369 (obsolete NCT alias)
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Depression; Lung Cancer
Keywords: depression; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Depression; Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Counseling; Psychiatric Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Arm I (control) (Experimental): Arm I (control): Patients complete screening questionnaires about their mood and experience with lung cancer once before and once after a visit with their physician. Neither the patient nor physician receives the screening results before the visit.
  Interventions: Other: counseling intervention; Other: screening questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: psychosocial assessment and care
- Arm II (Experimental): Arm II: Patients complete screening questionnaires as in arm I. Only the patient receives the screening results before their visit with the physician; the physician remains blinded to the results.
  Interventions: Other: counseling intervention; Other: screening questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: psychosocial assessment and care
- Arm III (Experimental): Arm III: Patients complete screening questionnaires as in arm I. Only the physician receives the screening results before their visit with the patient; the patient remains blinded to the results.
  Interventions: Other: counseling intervention; Other: screening questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: psychosocial assessment and care
- Arm IV (Experimental): Arm IV: Patients complete screening questionnaires as in arm I. Both physician and patient receive the screening results before the visit.
  All patients and physicians are notified of the screening results before the patient leaves the clinic. All patients are offered supportive counseling.
  Interventions: Other: counseling intervention; Other: screening questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: psychosocial assessment and care

INTERVENTIONS:
Other: counseling intervention
Other: screening questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Screening tests may help doctors find depression in patients with lung cancer, allow doctors to recommend treatment for depression, and improve the patient's quality of life.

PURPOSE: This randomized clinical trial is studying how well depression screening works when the results are or are not shared with patients with lung cancer and their doctor.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the impact of depression screening in patients with lung cancer when the results of the screening are made available to the patient, the physician, both, or neither on detection of depression, provision of depression treatment recommendations, and the quality of the doctor-patient interaction from the patient's perspective.

Secondary

* Determine psychological and demographic subsets for the impact of depression screening in these patients when the results of the screening are made available to the patient, the physician, both, or neither on the detection of depression, provision of depression treatment recommendations, and the quality of the doctor-patient interaction from the patient's perspective.

OUTLINE: This is a multicenter, randomized, double-blind, single-blind, factorial study. Patients are stratified according to participating center (Memorial Sloan-Kettering Cancer Center vs University of Kentucky Markey Cancer Center). Patients are randomized to 1 of 4 screening arms.

* Arm I (control): Patients complete screening questionnaires about their mood and experience with lung cancer once before and once after a visit with their physician. Neither the patient nor physician receives the screening results before the visit.
* Arm II: Patients complete screening questionnaires as in arm I. Only the patient receives the screening results before their visit with the physician; the physician remains blinded to the results.
* Arm III: Patients complete screening questionnaires as in arm I. Only the physician receives the screening results before their visit with the patient; the patient remains blinded to the results.
* Arm IV: Patients complete screening questionnaires as in arm I. Both physician and patient receive the screening results before the visit.

All patients and physicians are notified of the screening results before the patient leaves the clinic. All patients are offered supportive counseling.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of lung cancer
* Prescreening distress thermometer score > 3
* Zung Self-Rating Depression Scale (ZSDS) score ≥ 44

  * No ZSDS response indicating suicidality

PATIENT CHARACTERISTICS:

* Able to understand English
* No evidence of cognitive dysfunction that would impair giving consent

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2006-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of treatment recommendations for depression made as measured by checklist of recommendations for depression treatment | 2 years
Degree of patient satisfaction with interaction as measured by Medical Interview Satisfaction Scale | 2 years
Overall patient experience as measured by Patient Experience Questionnaire | 2 years

SECONDARY OUTCOMES:
Psychological and demographic subsets of patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William Breitbart, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Memorial Sloan-Kettering Cancer Center, New York, New York